CLINICAL TRIAL: NCT05312060
Title: Pneumatic Compression Versus Anti-thromboembolic Exercises: Effects on Edema of the Lower Limbs and the Outcomes of Patients Undergoing Total Hip Arthroplasty: Randomized Controlled Clinical Trial
Brief Title: Pneumatic Compression Versus Anti-thromboembolic Exercises for Patients Undergoing Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Luca Marin (Other)
Responsible Party: Sponsor-Investigator, Luca Marin, Principal Investigator, University of Pavia
Organization: University of Pavia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0014626/22
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Edema Leg
Keywords: Total hip arthroplasty; functional capabilities; Pneumatic compression; antithromboembolic exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumatic Compression (PC) (Experimental): The PC will undergo two daily 30-minute sessions of sequential pneumatic compression.
  Interventions: Device: PC Pneumatic compression
- Antithromboembolic exercises (AE) (Active Comparator): AE will perform two supervised antithromboembolic exercises sessions daily lasting 30 minutes.
  Interventions: Other: AE Antithromboembolic exercises

INTERVENTIONS:
Device: PC Pneumatic compression — Pneumatic compression of the operated limb
  Other Names: I-Press®, I-Tech Medical Division, Martellago, Italy
  Arms: Pneumatic Compression (PC)
Other: AE Antithromboembolic exercises — Exercises for the edema
  Arms: Antithromboembolic exercises (AE)

SUMMARY:
This study is a randomized controlled trial, with two parallel arms. The open-label study will be conducted in accordance with the helsinky statement and good clinical practice standards.

The main objective is to compare the reduction of postoperative edema following Total Hip Arthroplasty (THA) between patients undergoing postoperative treatment with pneumatic compression (PC, experimental group) and patients undergoing postoperative treatment with antithromboembolic exercises. (AE, control group). We also aim to compare the pre-post treatment variations of joint function measurements (joint excursion), referred pain and functional capabilities.

48 patients will meet the criteria listed below will be recruited.

Inclusion criteria:

* total hip arthroplasty under election regime
* aged between 50 and 80 at the time of recruitment, both sexes.

Exclusion criteria:

* obesity (BMI> 30);
* other orthopedic or neurological pathologies that modify walking ability;
* pathologies that modify balance (neurological and / or vestibular);
* contraindications to the use of the medical equipment used in the study;
* inability to understand and sign informed consent. Participants will be assigned, through a block randomization, to one of the two study groups: experimental group will undergo pneumatic compression treatment (PC), control group will perform antithromboembolic exercises (AE).

For both, the treatment will last 10 working days, starting from the first post surgery day (T0). The PC will undergo two daily 30-minute sessions of sequential pneumatic compression (I-Press®, I-Tech Medical Division, Martellago, Italy) while AE will perform two supervised antithromboembolic exercises sessions daily lasting 30 minutes. All participants will carry out the antithrombotic prophylaxis in use at the department of orthopedics: drug therapy, graduated compression stocking and indirect electrostimulation (T-One Rehab®, I-Tech Medical Division, Martellago, Italy).

Assessments of edema, joint range of motion, pain and functional capabilities will be made at T0 and at the end of the treatment (T1).

DETAILED DESCRIPTION:
This study is a randomized controlled trial, with two parallel arms. The open-label study will be conducted in accordance with the helsinky statement and good clinical practice standards.

To compare the reduction of postoperative edema following Total Hip Arthroplasty (THA) between patients undergoing postoperative treatment with pneumatic compression (PC, experimental group) and patients undergoing postoperative treatment with antithromboembolic exercises. (AE, control group). We also aim to compare the pre-post treatment variations of joint function measurements (joint excursion), referred pain and functional capabilities.

48 patients will be recruited at the Department of Orthopedic Surgery of the City of Pavia, University Hospital.

Participants will be assigned, through a block randomization, to one of the two study groups: experimental group will undergo pneumatic compression treatment (PC), control group will perform antithromboembolic exercises (AE). For both, the treatment will last 10 working days, starting from the first post surgery day (T0). The PC will undergo two daily 30-minute sessions of sequential pneumatic compression (I-Press®, I-Tech Medical Division, Martellago, Italy) while AE will perform two supervised antithromboembolic exercises sessions daily lasting 30 minutes. All participants will carry out the antithrombotic prophylaxis in use at the department of orthopedics: drug therapy, graduated compression stocking and indirect electrostimulation (T-One Rehab®, I-Tech Medical Division, Martellago, Italy).

At T0 and at the end of the treatment (T1) the following assessments of the operated limb will be carried out:

* circumference of the distal third of the thigh
* circumference of the proximal third of the leg
* range of motion of the knee flexion
* range of motion of the ankle dorsiflexion

The following assessments will also be carried out:

* perceived pain, with the Numeric Rating Scale of Pain (NRS)
* functional capability, with 20 m walk test (20 m). Walking autonomy will be carried out at T1 with the 6 minutes walking test (6MWT).

STATISTICAL ANALYSIS Quantitative variables will be described with mean and standard deviation if normally distributed, with median and interquartile range if not normally distributed.

Categorical variables will be expressed with counts and percentages. Continuous variables will be compared between the two groups with Student's t test or with the analogous non-parametric Mann-Whitney test, considering the normality of the distribution (evaluated with graphical methods or with the Shapiro-Wilk test).

Possible associations between categorical variables will be evaluated with Pearson's chi-square test or with Fisher's exact test.

All tests will be two-tailed; the level of significance is set at alpha 0.05 (statistical significance if p value <0.05).

ELIGIBILITY:
Inclusion Criteria:

* total hip arthroplasty, scheduled surgery
* aged between 50 and 80 at the time of recruitment

Exclusion Criteria:

* obesity (BMI> 30);
* other orthopedic or neurological pathologies that modify walking ability;
* pathologies that modify balance (neurological and / or vestibular);
* contraindications to the use of the medical equipment used in the study;
* inability to understand and sign informed consent.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Operated limb edema | Ten days
  circumference of the distal third of the thigh
  * circumference of the proximal third of the leg circumference of the distal third of the thigh
  * circumference of the proximal third of the leg thigh and leg circumference

SECONDARY OUTCOMES:
Perceived Pain | Ten days
  Perceived pain, assessed with Numeric Rating Scale. Where 0 is no pain and 10 is the maximum pain felt
Functional capability | Ten Days
  Walking capability, assessed with 20 meters walking test
Operated lower limb range of motion | Ten Days
  Knee and ankle range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marin, PhD, Principal Investigator — University fo Pavia
Locations (1):
- Istituto di Cura Città di Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santana DC, Emara AK, Orr MN, Klika AK, Higuera CA, Krebs VE, Molloy RM, Piuzzi NS. An Update on Venous Thromboembolism Rates and Prophylaxis in Hip and Knee Arthroplasty in 2020. Medicina (Kaunas). 2020 Aug 19;56(9):416. doi: 10.3390/medicina56090416. PMID 32824931
- [Background] O'Reilly RF, Burgess IA, Zicat B. The prevalence of venous thromboembolism after hip and knee replacement surgery. Med J Aust. 2005 Feb 21;182(4):154-9. doi: 10.5694/j.1326-5377.2005.tb06643.x. PMID 15720169
- [Background] Williams KJ, Ravikumar R, Gaweesh AS, Moore HM, Lifsitz AD, Lane TR, Shalhoub J, Babber A, Davies AH. A Review of the Evidence to Support Neuromuscular Electrical Stimulation in the Prevention and Management of Venous Disease. Adv Exp Med Biol. 2017;906:377-386. doi: 10.1007/5584_2016_128. PMID 27620314
- [Background] Westrich GH, Specht LM, Sharrock NE, Sculco TP, Salvati EA, Pellicci PM, Trombley JF, Peterson M. Pneumatic compression hemodynamics in total hip arthroplasty. Clin Orthop Relat Res. 2000 Mar;(372):180-91. doi: 10.1097/00003086-200003000-00020. PMID 10738427
- [Background] Berliner JL, Ortiz PA, Lee YY, Miller TT, Westrich GH. Venous Hemodynamics After Total Hip Arthroplasty: A Comparison Between Portable vs Stationary Pneumatic Compression Devices and the Effect of Body Position. J Arthroplasty. 2018 Jan;33(1):162-166. doi: 10.1016/j.arth.2017.08.005. Epub 2017 Aug 24. PMID 28927565
- [Background] Pitto RP, Hamer H, Kuhle JW, Radespiel-Troger M, Pietsch M. [Hemodynamics of the lower extremity with pneumatic foot compression. Effect on leg position]. Biomed Tech (Berl). 2001 May;46(5):124-8. doi: 10.1515/bmte.2001.46.5.124. German. PMID 11413908
- [Background] Pitto RP, Young S. Foot pumps without graduated compression stockings for prevention of deep-vein thrombosis in total joint replacement: efficacy, safety and patient compliance. A comparative, prospective clinical trial. Int Orthop. 2008 Jun;32(3):331-6. doi: 10.1007/s00264-007-0326-9. Epub 2007 Feb 15. PMID 17653546
- [Background] Fujisawa M, Naito M, Asayama I, Kambe T, Koga K. Effect of calf-thigh intermittent pneumatic compression device after total hip arthroplasty: comparative analysis with plantar compression on the effectiveness of reducing thrombogenesis and leg swelling. J Orthop Sci. 2003;8(6):807-11. doi: 10.1007/s00776-003-0706-y. PMID 14648269
- [Background] Zhao JM, He ML, Xiao ZM, Li TS, Wu H, Jiang H. Different types of intermittent pneumatic compression devices for preventing venous thromboembolism in patients after total hip replacement. Cochrane Database Syst Rev. 2014 Dec 22;2014(12):CD009543. doi: 10.1002/14651858.CD009543.pub3. PMID 25528992
- [Background] Kakkos SK, Caprini JA, Geroulakos G, Nicolaides AN, Stansby G, Reddy DJ, Ntouvas I. Combined intermittent pneumatic leg compression and pharmacological prophylaxis for prevention of venous thromboembolism. Cochrane Database Syst Rev. 2016 Sep 7;9(9):CD005258. doi: 10.1002/14651858.CD005258.pub3. PMID 27600864
- See also: Declaration of Helsinki — http://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects